CLINICAL TRIAL: NCT02676414
Title: Validation of the Hypertension Education Program of the German Hypertension League (DHL©) "My Blood Pressure - OK!"
Brief Title: Validation of a Hypertension Education Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Reinhold Kreutz, Professor, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DHL-HEP1
Record Dates: First submitted 2016-02-04; First posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Arterial Hypertension
MeSH Terms: conditions — Hypertension

ARMS (2):
- Education program (Other): Group of patients participating in the interactive hypertension education program of the DHL© "My blood pressure - OK!"
  Interventions: Behavioral: Interactive hypertension education program of the DHL©
- Controls (No Intervention): Group of patients not participating in the interactive hypertension education program of the DHL© "My blood pressure - OK!" ("usual care")

INTERVENTIONS:
Behavioral: Interactive hypertension education program of the DHL©
  Arms: Education program

SUMMARY:
The primary purpose of this study is to assess the effect of participating in the interactive hypertension education program of the German Hypertension League (DHL©) "My blood pressure - OK!" on office systolic blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* > 21 years of age
* Primary arterial hypertension
* Office blood pressure between 140/90 mmHg and 160/100 mmHg

Exclusion Criteria:

* Participation in another clinical study
* Unstable clinical condition
* Secondary arterial hypertension
* Dementia
* Major disability (modified Rankin-Scale > 4)
* Severe chronic kidney disease (serum creatinine > 2.0 mg/dL or estimated glomerular filtration rate < 40 ml/min/1.73m2)
* Liver disease including history of hepatic encephalopathy, esophageal varices or portacaval shunt
* History of gastrointestinal operation or disease with a potential influence on drug absorption
* Allergy or other contraindications against drugs given during the study
* History of non-compliance

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Office systolic blood pressure (mmHg) | 6 months

SECONDARY OUTCOMES:
Office diastolic blood pressure (mmHg) | 6 months
Self-measured systolic and diastolic blood pressure (mmHg) | 6 months
24-hour ambulatory blood pressure monitoring (mmHg) | 6 months
Body Mass Index (kg per m2) | 6 months
Physical activity (hours per week) | 6 months
Alcohol consumption (drinks per week) | 6 months
Quality of life based on the Quality of Life Questionnaire "The Short Form 36 Health Survey" | 6 months
Knowledge regarding arterial hypertension based on the DHL© Questionnaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Reinhold Kreutz, Professor, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Herz- und Diabeteszentrum Ruhr-Universität Bochum, Bad Oeynhausen, North Rhine-Westphalia, Germany